CLINICAL TRIAL: NCT06280118
Title: The Effect of Fatigue Caused by Search and Rescue Efforts in the Debris on the Quality of Cardiopulmonary Resuscitation: A Randomized Controlled Trial
Brief Title: The Effect of Fatigue on CPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Kadir Cavus, Lecturer (Phd-c), Artvin Coruh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EFCPR008
Record Dates: First submitted 2024-01-26; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Resuscitation
Keywords: Earthquake, debris, compression, ventilation, fatigue
MeSH Terms: conditions — Respiratory Aspiration; Fatigue

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pre-test (Control group) (No Intervention)
- Post test (Control group) (No Intervention)
- Pre test (experimental group) (No Intervention)
- Post test (experimental group) (Experimental)
  Interventions: Other: Fatigue

INTERVENTIONS:
Other: Fatigue — Fatigue was created in the participants by rehearsing the process of removing and transporting earthquake victims from the rubble through the prepared track.
  Arms: Post test (experimental group)

SUMMARY:
Background: This study, in contrast to the previous studies, generated a scenario of fatigue in an earthquake scenario and aimed to measure the effect of fatigue on the quality of cardiopulmonary resuscitation (CPR) performed by paramedics in a debris course.

Methods: The study was designed as a randomized controlled trial. The sample, consisting of 84 paramedic students, was randomly assigned as 42 control and 42 experimental groups. Fatigue was created in the participants by rehearsing the process of removing and transporting earthquake victims from the rubble through the prepared track. A personal information form and a CPR measurement form were used to obtain the data. The simulator was used to evaluate the accuracy of CPR. The collected data were analysed with the statistical program.

DETAILED DESCRIPTION:
Introduction Cardiopulmonary Arrest (CPA) is among the leading cause of death worldwide. Each year, 375,000 people are reported to die in Europe and 250,000 in the United States due to CPA. Early diagnosis of arrest and Cardiopulmonary Resuscitation is life-saving. However, earthquakes, one of the deadliest disasters, are among the most challenging situations that people around the world have to face. The rate of rescue of survivors from earthquake or collapsed structures is reported to decrease by 50% following 24 hours. Therefore, the first 72 hours are crucial for search and rescue operations in disasters. In earthquakes, while some of the disaster victims experience arrest at the scene due to trauma, others experience arrest in early or late periods depending on the injury site and localization. Thus, search and rescue operations should be initiated quickly, effectively and swiftly in disaster areas. Properly and efficiently administered CPR is among the most crucial life-saving emergency medical care methods. In Turkey, paramedics are also deployed to National Medical Rescue Team (NMRT) units to support search and rescue activities and provide emergency medical care. Paramedics have difficulties in maintaining chest compressions in arrest cases, especially in challenging cases in tight spaces outside the hospital. Since chest compressions are considered the essential element of CPR, their quality is thought to be affected under harsh conditions. 2015 International Liaison Committee on Resuscitation (ILCOR) recommended the compression depth as 5-6 cm and stated that 1/3 of the sternum should be compressed owing to the body mass differences of the rescuers. However, effective CPR depends on many parameters such as the number of rescuers, elapsed time, physical characteristics and muscle strength of the rescuer, high level of fitness, fatigue, weight of the rescuer, physical fitness, having a higher maximum oxygen consumption, position of the rescuer, difficult and confined space rescues. This study aimed in this context, to measure the effects of fatigue on CPR using high-quality simulators.

ELIGIBILITY:
Inclusion Criteria:

* Being a paramedic student.
* Having taken a resuscitation course.

Exclusion Criteria:

* None

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The groups were arranged by randomization with two female and one male participants.
Enrollment: 84 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
Correct number of ventilations | 120 second
  The number of ventilations applied correctly will be measured in the pre-test and post-tests.
Correct number of compression | 120 second
  The number of compressions applied in the correct way will be measured in the pre-test and post-test.

SECONDARY OUTCOMES:
CPR duration | 120 second
  CPR times applied in the pre-test and post-test will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Oğuzhan Tiryaki, Expert Nursing, Principal Investigator — Artvin State Hospital; Elif Tiryaki, Lecturer, Principal Investigator — Artvin Çoruh University; Suat Çelik, Lecturer, Principal Investigator — Artvin Çoruh University; Hüseyin Bora Saçar, Lecturer, Principal Investigator — Artvin Çoruh University
Locations (1):
- Resuscitation simulation laboratory of Artvin Çoruh University Health Services Vocational School, Artvin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pan DF, Li ZJ, Ji XZ, Yang LT, Liang PF. Video-assisted bystander cardiopulmonary resuscitation improves the quality of chest compressions during simulated cardiac arrests: A systemic review and meta-analysis. World J Clin Cases. 2022 Nov 6;10(31):11442-11453. doi: 10.12998/wjcc.v10.i31.11442. PMID 36387811
- [Background] Kleinman ME, Brennan EE, Goldberger ZD, Swor RA, Terry M, Bobrow BJ, Gazmuri RJ, Travers AH, Rea T. Part 5: Adult Basic Life Support and Cardiopulmonary Resuscitation Quality: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S414-35. doi: 10.1161/CIR.0000000000000259. No abstract available. PMID 26472993